CLINICAL TRIAL: NCT04246216
Title: Ultrasound-Guided Percutaneous Electrical Nerve Stimulation of the Median Nerve for Carpal Tunnel Syndrome
Brief Title: Percutaneous Electrical Nerve Stimulation for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Full proffessor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC0209201911819
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Electrical Nerve Stimulation (Experimental): The experimental group will receive 3 sessions (once per week) of ultrasound-guided Percutaneous Electrical Nerve Stimulation targeted the median nerve. Once the median nerve is ultrasound identified, the needles will be left in situ at the identified points connected to an electrostimulator (ES-160 ITO co.) applying a biphasic continuous waveform, at low frequency (2 Hz)19 and with 250 microseconds pulse duration for 30mins.
  Interventions: Procedure: Percutaneous Electrical Nerve Stimulation
- Surgery (Active Comparator): The surgical group will receive a surgical procedure consisting of the decompression and release of the median nerve at the carpal tunnel performed by an experienced surgeon according to standardized protocols.
  Interventions: Procedure: Endoscopic surgery of the carpal tunnel

INTERVENTIONS:
Procedure: Percutaneous Electrical Nerve Stimulation — Experimental: Percutaneous Electrical Nerve Stimulation The experimental group will receive 3 sessions (once per week) of ultrasound-guided Percutaneous Electrical Nerve Stimulation targeted the median nerve. Once the median nerve is ultrasound identified, the needles will be left in situ at the identified points connected to an electrostimulator (ES-160 ITO co.) applying a biphasic continuous waveform, at low frequency (2 Hz)19 and with 250 microseconds pulse duration for 30mins.
  Arms: Percutaneous Electrical Nerve Stimulation
Procedure: Endoscopic surgery of the carpal tunnel — The surgical group will receive a surgical procedure consisting of the decompression and release of the median nerve at the carpal tunnel performed by an experienced surgeon according to standardized protocols.
  Arms: Surgery

SUMMARY:
There is evidence supporting that physical therapy interventions can be effective for the management of patients with CTS. No consensus on the best approach exist. It seems clear that the median nerve is affected in several ways (compression, inflammation, excursion) in carpal tunnel syndrome. Percutaneous Electrical Nerve Stimulation is a treatment approach consisting of the application of an electrical current throughout needling filaments placed close to the nerve, in this case the median nerve. The purpose of this clinical trial is to compare changes in function, symptom severity and the intensity of pain after the application of Percutaneous Electrical Nerve Stimulation vs. endoscopic surgery in women with CTS at short- and long-term follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* pain and paresthesia in the median nerve distribution
* positive Tinel sign,
* positive Phalen sign,
* symptoms had to have persisted for at least 6 months
* deficits of sensory and motor median nerve conduction according to guidelines of the American Association of Electrodiagnosis, American Academy of Neurology, and the American Physical Medicine and Rehabilitation Academy

Exclusion Criteria:

* any sensory/motor deficit related to the ulnar or radial nerve;
* older than 65 years of age;
* previous surgical intervention, steroid injections or physical therapy intervention
* multiple diagnoses of the upper extremity (eg, cervical radiculopathy);
* history of neck, shoulder, or upper limb trauma (whiplash);
* history of any systemic disease causing CTS (eg, diabetes mellitus, thyroid disease);
* history of other systemic conditions (eg, rheumatoid arthritis, fibromyalgia);
* pregnancy;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity between baseline and follow-up periods | Baseline and 1, 3, 6 and 12 months after the intervention.
  An 11-point Numerical Pain Rating Scale (NPRS, 0: no pain - 10: maximum pain) will be used to assess the patients' current level of hand pain and the worst and lowest level of pain experienced in the preceding week.

SECONDARY OUTCOMES:
Changes in hand function between baseline and follow-up periods | Baseline and 1, 3, 6 and 12 months after the intervention.
  The Spanish version of the Boston Carpal Tunnel Questionnaire (BCTQ) will be used to assess function. This questionnaire evaluates 2 domains: 1) the functional status scale assesses ability to perform 8 common hand-related tasks; and, 2) the symptom severity scale includes 11 items assessing pain severity, numbness, and weakness at night and during the day. Each question is answered on a 5-point scale (1: no complaint; 5: severe complaint), with higher scores indicating greater severity.
Changes in severity between baseline and follow-up periods | Baseline and 1, 3, 6 and 12 months after the intervention.
  The Spanish version of the Boston Carpal Tunnel Questionnaire (BCTQ) will be used to assess function. This questionnaire evaluates 2 domains: 1) the functional status scale assesses ability to perform 8 common hand-related tasks; and, 2) the symptom severity scale includes 11 items assessing pain severity, numbness, and weakness at night and during the day. Each question is answered on a 5-point scale (1: no complaint; 5: severe complaint), with higher scores indicating greater severity.
Changes in patient self-perceived improvement between baseline and follow-up periods | Baseline and 1, 3, 6 and 12 months after the intervention.
  . Subjects self-perceived improvement will be assessed using a Global Rating of Change (GROC) which consists of a 15-point scale ranging from -7 (a very great deal worse) to +7 (a very great deal better). It has been reported that scores of +4 and +5 are indicative of moderate changes in patient status, whereas scores of +6 and +7 indicate large changes in the status of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: César Fernández-de-las-Peñas, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- César Fernández-de-las-Peñas, Alcorcón, Alcorcon, Madrid, Spain

REFERENCES:
- [Derived] Fernandez-de-Las-Penas C, Ortega-Santiago R, De-la-Llave-Rincon AI, Cleland JA, Pareja JA, Fahandezh-Saddi-Diaz H, Arias-Buria JL. Ultrasound-guided percutaneous electrical nerve stimulation versus surgery for women with unilateral carpal tunnel syndrome: A randomized parallel-group trial. Eur J Pain. 2023 Aug;27(7):860-870. doi: 10.1002/ejp.2117. Epub 2023 Apr 7. PMID 36987682